CLINICAL TRIAL: NCT01390779
Title: Efficacy of 24-hour Intraocular Pressure Fluctuation Recording With the SENSIMED Triggerfish Contact Lens Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10/09
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2013-12

CONDITIONS: Primary Open Angle Glaucoma; Healthy Subjects
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SENSIMED Triggerfish (Experimental): All subjects enrolled in the trial were housed in a sleep laboratory for 24 hours, during which they underwent SENSIMED Triggerfish recording on one randomly selected eye.
  Interventions: Device: SENSIMED Triggerfish

INTERVENTIONS:
Device: SENSIMED Triggerfish — Contact lens-based device intended to continuously record the timing of relative changes in IOP for up to 24 hours

SUMMARY:
The objectives of this study are to assess the safety and effectiveness of the SENSIMED Triggerfish® (TF) device in continuous recording of relative fluctuation in intraocular pressure (IOP). Safety will be assessed by recording of AEs during the 24 hours of continuous TF recording.

TF efficacy will be evaluated by demonstrating TF ability to detect:

1. The known phenomenon of increase in IOP when moving from waking state to going to bed, as reflected in pneumotonometer measurements
2. Ocular Pulse frequency relative to direct measurement of Heart Rate (HR).

A screening visit and one 24-hour IOP fluctuation recording session are planned for each patient. IOP fluctuation recording sessions will be carried out in a sleep unit. An ophthalmological examination of the eyes will be done at screening and prior to and following the device recording.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent for the investigation
* Diagnosis of primary open angle glaucoma (POAG), including normal tension glaucoma, or healthy subjects, including subjects with ocular hypertension for whom no evidence or suspicion of structural or functional glaucomatous damage exists
* No anti-glaucomatous drug treatment or washed-out for 4 weeks
* IOP symmetry of +/- 3 mmHg between fellow eyes
* Age 18-80 years
* Not more than 4 diopters spherical equivalent on both eyes
* Not more than 2 diopters cylinder equivalent on both eyes

Exclusion Criteria:

* Patients who have had ocular surgery within the last 3 months.
* Corneal or conjunctival abnormality hindering contact lens adaptation
* Wear of full frame metallic glasses during SENSIMED Triggerfish® monitoring
* Severe dry eye
* Secondary forms of open angle glaucoma (OAG)
* Allergy to corneal anesthetic
* Patients with contraindications for silicone contact lens wear
* Patients not able to understand the character and individual consequences of the investigation
* Simultaneous participation in other clinical research

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John HK Liu, PhD, Principal Investigator — UCSD
Locations (1):
- UCSD, San Diego, California, United States

REFERENCES:
- [Derived] Mansouri K, Weinreb RN, Liu JH. Efficacy of a contact lens sensor for monitoring 24-h intraocular pressure related patterns. PLoS One. 2015 May 5;10(5):e0125530. doi: 10.1371/journal.pone.0125530. eCollection 2015. PMID 25942434

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from July 2011 to May 2012, from medical clinic and investigator's patient database.
Pre-assignment Details: Regular sleep cycle in the week preceding the study.
Groups:
- SENSIMED Triggerfish: All subjects enrolled in the trial were housed in a sleep laboratory for 24 hours, during which they underwent SENSIMED Triggerfish recording on one randomly selected eye.
  Parallel IOP measurements were taken using pneumatonometry on the eye contralateral to the SENSIMED Triggerfish eye before and after sleep onset. During sleep heart rate measurements were collected at specified time points.
Period: Overall Study
Arm/Group | SENSIMED Triggerfish
Started | 33
Completed | 32
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | SENSIMED Triggerfish
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: SENSIMED Triggerfish Efficacy
Description: Investigate the device's capacity to detect changes in IOP from wake to sleep, defined as a significantly positive slope on the SENSIMED Triggerfish recording (obtained on one eye in each subject), based on the established phenomenon that IOP increases from waking to sleep hours. The IOP from wake to sleep was measured in the eye contralateral to that of SENSIMED Triggerfish using pneumatonomtery. Subjects were included in the primary analysis if a difference in IOP of at least 3 mmHg was detected from wake to sleep.
  One subject was excluded from the analysis due to the absence of a 3-mmHg difference in IOP from wake to sleep. Two subjects were excluded since they had less than 80% of expected SENSIMED Triggerfish data. One subject was excluded from the analysis due to an invalid SENSIMED Triggerfish recording.
Time Frame: from 1 hour before sleep to 1 hour after sleep
Population: Subjects were included in this analysis if the difference in IOP from wake to sleep was at least 3 mmHg, as determined using pneumatonometry on the eye contralateral to that of SENSIMED Triggerfish, and if the SENSIMED Triggerfish recording contained at least 80% of the expected data points.
Measure: Mean (Standard Deviation); unit: mV/h
Arm/Group | SENSIMED Triggerfish
Number analyzed (Participants) | 29
mV/h | 56.9 (40.5)

2. Primary Outcome: SENSIMED Triggerfish Efficacy
Description: Device's ability to detect ocular pulse frequency concurrent to heart rate, defined as the number of SENSIMED Triggerfish recording intervals showing oscillation at a frequency matching that of heart rate +/- 15%. In absence of eye blinks during sleep, an oscillating pattern is recorded. The frequency of oscillation was determined by independent reviewers for selected SENSIMED Triggerfish 30-second recording intervals for which simultaneous or close to simultaneous heart rate data was recorded. Intervals for which the oscillation frequency on SENSIMED Triggerfish pattern matched heart rate +/- 15% (tolerance due to noise caused by eye and lid movements) were considered accurate. The percentage of accurate intervals was calculated and expected to be at least 75%.
Time Frame: in selected 30-second SENSIMED Triggerfish recording intervals during sleep
Population: One subject was excluded from the analysis due to the absence of a 3-mmHg difference in IOP from wake to sleep. Two subjects were excluded since they had less than 80% of expected SENSIMED Triggerfish data. One subject was excluded from the analysis due to an invalid SENSIMED Triggerfish recording.
Measure: Number (95% Confidence Interval); unit: % of accurate recording intervals
Arm/Group | SENSIMED Triggerfish
Number analyzed (Participants) | 29
% of accurate recording intervals | 86.5 [75 to 93.2]

ADVERSE EVENTS:
Arm/Group | SENSIMED Triggerfish
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 15/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SENSIMED Triggerfish (N=33)
ocular hyperemia (Eye disorders) | 8 (8)
punctate keratitis (Eye disorders) | 7 (7)
eye pressure mark (Eye disorders) | 5 (5)
vision blurred (Eye disorders) | 1 (1)
eyelid edema (Eye disorders) | 1 (1)
corneal disorder (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No